CLINICAL TRIAL: NCT04611581
Title: Objective Assessment of Behavioural Disorders in Parkinson's Disease
Brief Title: Objective Assessment of Behavioural Disorders in PD
Acronym: TECHNO-PARK
Status: Active, not recruiting | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: University of Bern (Other); University of Oxford (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-01777
Record Dates: First submitted 2020-10-15; First posted 2020-11-02 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: Parkinson's Disease; Non-motor Symptoms
Keywords: Parkinson's Disease; Non-motor symptoms; Assessment of non-motor symptoms; Sensor monitoring; Behavioural disorders; Deep Brain Stimulation; Apathy; Impulse Control Disorder
MeSH Terms: conditions — Parkinson Disease; Mental Disorders; Lethargy; Disruptive, Impulse Control, and Conduct Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- PD patients with apathy: PD patients with apathy according to the diagnostic criteria by Robert et al. 2018
- PD patients with impulse control disorder: PD patients with a) at least one item >2 or b) at least two items >1 on the hyperdopaminergic subscale of the Ardouin Scale of Behaviour in Parkinson's Disease
- PD patients without any relevant neuropsychiatric symptoms: PD patients with a score <2 on each item of the Ardouin Scale of Behaviour in Parkinson's Disease

SUMMARY:
The aim of this project is to measure behavioural disorders in Parkinson's disease (PD) patients in a more objective way, in order to facilitate the detection of those symptoms and improve the treatment of non-motor symptoms in Parkinson's disease.

DETAILED DESCRIPTION:
Apathy and impulse control disorders (ICDs) are frequent non-motor symptoms of PD and negatively affect the quality of life of patients. Although healthcare professionals have begun to understand the extent of the problem faced by those suffering apathy or ICDs, accurate diagnosis is still difficult, as behavioural symptoms are often multidimensional, develop gradually over the course of months and clinical staff have to rely on the self-report of the patient or the report of a family member to assess them. To overcome this issue, the investigators aim to use information and communication technologies to measure apathy and hyperdopaminergic behaviours in PD patients with STN-DBS in an objective way, with the ultimate goal of improving the management of PD patients with STN-DBS.

To do so, the investigators will use three computer-based tasks that measure effort-based decision making and emotion processing in PD patients, and assess motor, cognitive and neuropsychiatric symptoms in parallel with scales and tests. In some select patients, motor symptoms and activity patterns will be monitored with an in-home sensor system before and after deep brain stimulation STN-DBS, and the above mentioned procedures will be repeated 4 months after STN-DBS.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Parkinson's disease.
* (Planned) STN-DBS.
* Able to understand instructions and provide informed consent.
* Native speaking or proficient French or German
* Montreal Cognitive Assessment (MoCA) with score ≥ 22
* Ability to manipulate handheld dynamometers

Exclusion Criteria:

* Disease affecting the brain other than Parkinson's disease
* Suffering from or diagnosed with ongoing psychiatric illnesses
* Severe somatic illnesses leading to reduced life expectancy
* Severe physical disability leading to impairment in basic functional activities
* Participation in a pharmacological study
* Inability to provide informed consent (legal guardianship)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with idiopathic Parkinson's disease, treated at the movement disorders clinic in the University Hospital of Bern, Switzerland.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Performance in an effort-based decision making task (Apple Tree Paradigm) | Visit 1 (only visit for most patients; for DBS patients 1-3 months before DBS-surgery)
  Decision (yes/no)
Performance in an effort-based decision making task (Apple Tree Paradigm) | Visit 2 (only for DBS patients; 4-6 months after DBS-surgery)
  Decision (yes/no)
Performance in an emotion processing task | Visit 1 (only visit for most patients; for DBS patients 1-3 months before DBS-surgery)
  Pupil diameter (in mm)
Performance in an emotion processing task | Visit 2 (only for DBS patients; 4-6 months after DBS-surgery)
  Pupil diameter (in mm)
Change in overall activity from Baseline to 4 months after DBS-surgery | In-home sensor measurements will be collected from 1-3 months before DBS-surgery and 4 months after DBS-surgery
  Changes in overall activity patterns related to motivated behaviours (measured in minutes per day) will be deducted from collected from in-home sensor data using signal processing and machine learning algorithms

CONTACTS AND LOCATIONS:
Overall Officials: Paul Krack, MD, Principal Investigator — Insel Gruppe AG, University Hospital Bern
Locations (1):
- Insel Gruppe AG University Hospital of Bern, Bern, Switzerland